CLINICAL TRIAL: NCT04884191
Title: Phase 2 Study: An Open-Label, Randomized, Phase 2 Dose-Finding Study of Pacritinib in Patients With Primary Myelofibrosis, Post-Polycythemia Vera Myelofibrosis, or Post- Essential Thrombocythemia Myelofibrosis Previously Treated With Ruxolitinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAC203
Record Dates: First submitted 2021-05-10; First posted 2021-05-12 (Actual); Results first posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Primary Myelofibrosis; Post-Polycythemia Vera Myelofibrosis; Post- Essential Thrombocythemia Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pacritinib 100 mg QD (Experimental)
  Interventions: Drug: Pacritinib
- Pacritinib 100 mg BID (Experimental)
  Interventions: Drug: Pacritinib
- Pacritinib 200 mg BID (Experimental)
  Interventions: Drug: Pacritinib

INTERVENTIONS:
Drug: Pacritinib — Pacritinib

SUMMARY:
This was an open-label, randomized, dose-finding study in patients with primary or secondary MF (Dynamic International Prognostic Scoring System [DIPSS] risk score of Intermediate-1 to High-Risk) who were previously treated with ruxolitinib. The study was designed to support a pacritinib dosage selection decision with evaluation of 3 dosages.

ELIGIBILITY:
Inclusion Criteria:

1. PMF, PPV-MF, or PET-MF (as defined by Tefferi and Vardiman 2008)
2. DIPSS Intermediate-1, Intermediate -2, or High-risk (Passamonti et al 2010)
3. Prior ruxolitinib treatment with failure to benefit or intolerance as defined by at least one of the following:

   1. Treatment for ≥3 months with inadequate efficacy response defined as <10% SVR by MRI or <30% decrease from baseline in spleen length by physical examination or regrowth to these parameters following an initial response; and/or
   2. Treatment for ≥28 days complicated by either

   i. Development of a red blood cell (RBC) transfusion requirement (at least 2 units/month for 2 months) ii. National Cancer Institute (NCI) CTCAE grade ≥3 AEs of thrombocytopenia, anemia, hematoma, and/or hemorrhage while being treated with a dosage of <20 mg BID
4. Palpable splenomegaly ≥5 cm below the lower costal margin (LCM) in the midclavicular line as assessed by physical examination
5. TSS of ≥10 on the MPN-SAF TSS 2.0 or patients with a single symptom score of ≥5 or 2 symptoms of ≥3, including only the symptoms of left upper quadrant pain, bone pain, itching, or night sweats
6. Age ≥18 years old
7. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
8. Peripheral blast count of <10% throughout the Screening period
9. Absolute neutrophil count of >500/μL
10. Adequate liver and renal function, defined by liver transaminases (aspartate aminotransferase [AST]/serum glutamic-oxaloacetic transaminase [SGOT] and alanine aminotransferase [ALT]/serum glutamic-pyruvic transaminase [SGPT]), ≤3 × the upper limit of normal (ULN) (AST/ALT ≤5 × ULN, if transaminase elevation is related to MF), direct bilirubin ≤4× ULN, and creatinine ≤2.5 mg/dL
11. Adequate coagulation function, defined by prothrombin time (PT)/international normalized ratio (INR), partial thromboplastin time (PTT), or thrombin time (TT) of ≤1.5 × ULN
12. Left ventricular cardiac ejection fraction of ≥45% by echocardiogram or multigated acquisition (MUGA) scan
13. If fertile, willing to use effective birth control methods during the study
14. Willing to undergo and able to tolerate frequent MRI or CT scan assessments during the study
15. Able to understand and willing to complete symptom assessments using a PRO instrument
16. Provision of informed consent

Exclusion Criteria:

1. Life expectancy <6 months
2. Completed allogeneic stem cell transplant (allo-SCT) or are eligible for and willing to complete allo-SCT
3. History of splenectomy or planning to undergo splenectomy
4. Splenic irradiation within the last 6 months
5. Previously treated with pacritinib
6. Patients receiving high-dose ruxolitinib (more than 10 mg BID or 20 mg QD) who cannot tolerate tapering down ruxolitinib to 10 mg BID or less prior to the first dose of pacritinib
7. Treatment with anticoagulation or antiplatelet agents, except for aspirin dosages of ≤100 mg per day, within the last 2 weeks
8. Treatment with a strong CYP3A4 inhibitor or a strong cytochrome P450 inducer within the last 2 weeks
9. Treatment with medications that can prolong the QTc interval within the last 2 weeks
10. Treatment with an experimental therapy within the last 28 days
11. Significant recent bleeding history defined as NCI CTCAE grade ≥2 within the last 3 months, unless precipitated by an inciting event (eg, surgery, trauma, or injury)
12. Any history of CTCAE grade ≥2 non-dysrhythmia cardiac conditions within the last 6 months. Patients with asymptomatic grade 2 non-dysrhythmia cardiac conditions may be considered for inclusion, with the approval of the medical monitor, if stable and unlikely to affect patient safety.
13. New York Heart Association Class II, III, or IV congestive heart failure
14. Any history of CTCAE grade ≥2 cardiac dysrhythmias within the last 6 months. Patients with non-QTc CTCAE grade 2 cardiac dysrhythmias may be considered for inclusion, with the approval of the medical monitor, if the dysrhythmias are stable, asymptomatic, and unlikely to affect patient safety.
15. QTc prolongation >450 ms based on the mean of triplicate ECGs or other factors that increase the risk for QT interval prolongation (eg, heart failure, hypokalemia [defined as serum potassium <3.0 mEq/L that is persistent and refractory to correction], family history of long QT interval syndrome, or concomitant use of medications that may prolong QT interval)
16. Any active gastrointestinal or metabolic condition that could interfere with absorption of oral medication
17. Active or uncontrolled inflammatory or chronic functional bowel disorder such as Crohn's Disease, inflammatory bowel disease, chronic diarrhea, or constipation
18. Other malignancy within the last 3 years, other than curatively treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, organ-confined or treated nonmetastatic prostate cancer with negative prostate-specific antigen, in situ breast carcinoma after complete surgical resection, or superficial transitional cell bladder carcinoma
19. Uncontrolled intercurrent illness, including, but not limited to, ongoing active infection or psychiatric illness or social situation that, in the judgment of the treating physician, would limit compliance with study requirements
20. Known seropositivity for human immunodeficiency virus
21. Known active hepatitis A, B, or C virus infection
22. Women who are pregnant or lactating
23. Concurrent enrollment in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (62):
- United States (33):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - City of Hope, Duarte, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Stanford Cancer Institute, Stanford, California
  - Yale School of Medicine, New Haven, Connecticut
  - Medical Faculty Associates, Inc., Washington D.C., District of Columbia
  - Florida Cancer Specialists & Research Institute, Fort Myers, Florida
  - Florida Cancer Specialists & Research Institute, St. Petersburg, Florida
  - Florida Cancer Specialists & Research Institute, West Palm Beach, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - Saint Agnes Hospital, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University Hospital, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio School of Medicine, San Antonio, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- France (7):
  - CHU Hopital Sud, Amiens
  - Centre Hospitalier Regional Universitaire de Lille - Hopital Claude Huriez, Lille
  - CHU de Nimes - Hopital Universitaire Caremeau, Nîmes
  - Hôpital Saint-Louis, Paris
  - CHU Hopitaux de Bordeaux - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Toulouse- Hôpital Purpan, Toulouse
- Hungary (3):
  - SE AOK I. sx. Belgyogyaszati Klinika, Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
- Italy (3):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Istituto Scientifico Romagnolo per lo Studio e la Cura Dei Tumori, Meldola
  - ASST Monza - Ospedale San Gerardo, Monza
- South Korea (4):
  - Yeungnam University Medical Center, Daegu
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (4):
  - Hospital del Mar, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Clínica Universidad de Navarra, Pamplona
- Sweden (2):
  - Skane University Hospital Lund, Lund
  - Orebro University Hospital, Örebro
- United Kingdom (6):
  - Beatson West of Scotland Cancer Center, Glasgow
  - Barts Health NHS Trust - The Royal London Hospital, London
  - Guy's and St Thomas' NHS Foundation Trust - Guy's Hospital, London
  - Imperial College Healthcare NHS Trust - Hammersmith Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Trust - Churchill Hospital, Oxford

REFERENCES:
- [Derived] Verstovsek S, Mesa R, Talpaz M, Kiladjian JJ, Harrison CN, Oh ST, Vannucchi AM, Rampal R, Scott BL, Buckley SA, Craig AR, Roman-Torres K, Mascarenhas JO. Retrospective analysis of pacritinib in patients with myelofibrosis and severe thrombocytopenia. Haematologica. 2022 Jul 1;107(7):1599-1607. doi: 10.3324/haematol.2021.279415. PMID 34551507

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pacritinib 100 mg QD | Pacritinib 100 mg BID | Pacritinib 200 mg BID
Started | 55 | 55 | 55
Completed | 52 | 55 | 54
Not Completed | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pacritinib 100 mg QD | Pacritinib 100 mg BID | Pacritinib 200 mg BID | Total
Number analyzed (Participants) | 52 | 55 | 54 | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 11 | 16 | 43
  >=65 years | 36 | 44 | 38 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (8.8) | 68.9 (6.9) | 68.1 (8.76) | 68.7 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 26 | 22 | 69
  Male | 31 | 29 | 32 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 4 | 5
  White | 44 | 47 | 48 | 139
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 7 | 0 | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI not measured for all participants
  kg/m^2
    number analyzed (Participants) | 44 | 48 | 48 | 140
    (all) | 25.1 (3.79) | 27.2 (4.11) | 26.4 (5) | 26.3 (4.4)
ECOG PS [Number; unit: participants] — ECOG Performance Status 0 = Fully active, able to carry on all pre-disease performance without restriction
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. = Dead
  participants
    0 | 11 | 14 | 17 | 42
    1 | 32 | 29 | 29 | 90
    2 | 9 | 12 | 8 | 29

OUTCOME MEASURES:

1. Primary Outcome: Spleen Volume Reduction Response (≥ 35%)
Description: Number of patients achieving a ≥ 35% spleen volume reduction (SVR) as measured by magnetic resonance imaging (MRI, preferred) or computed tomography (CT) scans
Time Frame: From Baseline to Weeks 12 and 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pacritinib 100 mg QD | Pacritinib 100 mg BID | Pacritinib 200 mg BID
Number analyzed (Participants) | 52 | 55 | 54
Participants
  End of Week 12 | 0 | 2 | 2
  End of Week 24 | 0 | 1 | 5

2. Primary Outcome: Percent Change in Spleen Volume
Description: Percent change from baseline
Time Frame: From Baseline to Weeks 12 and 24
Population: The difference between the number of participants analyzed in Week 12 vs. Week 24 is the result of the number of participants that continued to complete the study. Participants that were not analyzed were withdrawn from the study for various reasons.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Pacritinib 100 mg QD | Pacritinib 100 mg BID | Pacritinib 200 mg BID
Number analyzed (Participants) | 38 | 43 | 43
percent change from baseline
  Week 12 | 3.19 (22.613) | 6.37 (31.110) | -3.60 (26.610)
  Week 24: number analyzed (Participants) | 26 | 26 | 27
  Week 24 | -2.43 (17.608) | 0.65 (20.589) | -11.30 (26.417)

3. Primary Outcome: Total Symptom Score Analysis
Description: Proportion of patients with ≥ 50% reduction in Total Symptom Score from baseline as assessed by the validated PRO instrument MPN-SAF TSS 2.0
Time Frame: From Baseline to Weeks 12 and 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pacritinib 100 mg QD | Pacritinib 100 mg BID | Pacritinib 200 mg BID
Number analyzed (Participants) | 52 | 55 | 54
Participants
  End of Week 12 | 1 | 1 | 2
  End of Week 24 | 2 | 0 | 2

4. Primary Outcome: Patient Global Impression Assessment
Description: Number of patients with improvement in PGIA. The Patient Global Impression Assessment questionnaire was completed at the end of Week 12 and end of Week 24. The scores were summarized by treatment group at each visit.
Time Frame: From Baseline to Weeks 12 and 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pacritinib 100 mg QD | Pacritinib 100 mg BID | Pacritinib 200 mg BID
Number analyzed (Participants) | 52 | 55 | 54
Participants
  Week 12 - Any Improved | 17 | 21 | 23
  Week 12 -No Change | 6 | 5 | 8
  Week 12 -Any Worse | 8 | 8 | 3
  Week 24 - Any Improved | 10 | 13 | 18
  Week 24 -No Change | 6 | 5 | 1
  Week 24 -Any Worse | 5 | 3 | 2

5. Secondary Outcome: Spleen Length Reduction
Description: Rate of reduction in spleen length from baseline
Time Frame: From Baseline to Weeks 24
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Pacritinib 100 mg QD | Pacritinib 100 mg BID | Pacritinib 200 mg BID
Number analyzed (Participants) | 24 | 25 | 27
cm | 12.42 (5.602) | 11.48 (6.501) | 11.63 (7.131)

6. Secondary Outcome: Frequency of RBC's or Platelet Transfusions
Description: Number of patients
Time Frame: At week 24
Measure: Mean (Standard Deviation); unit: transfusions/month
Arm/Group | Pacritinib 100 mg QD | Pacritinib 100 mg BID | Pacritinib 200 mg BID
Number analyzed (Participants) | 20 | 20 | 20
transfusions/month | 2.27 (2.987) | 1.18 (2.553) | 2.25 (2.345)

7. Secondary Outcome: Eastern Cooperative Oncology Group Performance Status
Description: 0 = Fully active, able to carry on all pre-disease performance without restriction
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. = Dead
Time Frame: At weeks 4, 12, 24, and 30 days post End-of-Treatment visit
Measure: Count of Participants; unit: Participants
Arm/Group | Pacritinib 100 mg QD | Pacritinib 100 mg BID | Pacritinib 200 mg BID
Number analyzed (Participants) | 52 | 55 | 54
Participants
  Week 4 - 0 | 10 | 11 | 13
  Week 4 - 1 | 28 | 27 | 31
  Week 4 - 2 | 9 | 16 | 8
  Week 4 - 3 | 2 | 0 | 0
  Week 4 - 4 | 0 | 0 | 0
  Week 4 - 5 | 0 | 0 | 0
  Week 12 - 0 | 11 | 9 | 14
  Week 12 - 1 | 20 | 23 | 19
  Week 12 - 2 | 8 | 10 | 8
  Week 12 - 3 | 1 | 1 | 2
  Week 12 - 4 | 0 | 0 | 0
  Week 12 - 5 | 0 | 0 | 0
  Week 24 - 0 | 10 | 6 | 10
  Week 24 - 1 | 12 | 15 | 12
  Week 24 - 2 | 4 | 5 | 6
  Week 24 - 3 | 0 | 0 | 0
  Week 24 - 4 | 0 | 0 | 0
  Week 24 - 5 | 0 | 0 | 0
  End of Treatment - 0 | 11 | 8 | 8
  End of Treatment - 1 | 19 | 23 | 22
  End of Treatment - 2 | 5 | 10 | 11
  End of Treatment - 3 | 1 | 1 | 2
  End of Treatment - 4 | 0 | 0 | 0
  End of Treatment - 5 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Randomization through 30 days post End-of-Treatment visit
Population: Patients with ≥ 1 TEAE
Measure: Count of Participants; unit: Participants
Arm/Group | Pacritinib 100 mg QD | Pacritinib 100 mg BID | Pacritinib 200 mg BID
Number analyzed (Participants) | 52 | 55 | 54
Participants | 49 | 51 | 54

ADVERSE EVENTS:
Time Frame: The end of assigned study drug + 30 days
Description: AEs analyzed in the Safety Population
Arm/Group | Pacritinib 100 mg QD | Pacritinib 100 mg BID | Pacritinib 200 mg BID
All-Cause Mortality (participants affected / at risk) | 6/52 | 4/55 | 5/54
Serious Adverse Events (participants affected / at risk) | 19/52 | 20/55 | 25/54
Other Adverse Events (participants affected / at risk) | 24/52 | 34/55 | 36/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pacritinib 100 mg QD (N=52) | Pacritinib 100 mg BID (N=55) | Pacritinib 200 mg BID (N=54)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 2 | 3
General physical health deterioration (General disorders) | 2 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 2 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 5
Cellulitis (Infections and infestations) | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 2
Tuberculosis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 2
Herpes oesophagitis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Delayed haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incorrect drug administration duration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 2
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Optic neuritis (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 2
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Renal mass (Renal and urinary disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung infiltration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 1
Vascular compression (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pacritinib 100 mg QD (N=52) | Pacritinib 100 mg BID (N=55) | Pacritinib 200 mg BID (N=54)
Diarrhoea (Gastrointestinal disorders) | 6 | 8 | 14
Nausea (Gastrointestinal disorders) | 7 | 7 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 5 | 9
Fatigue (General disorders) | 1 | 7 | 5
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 6
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 3
Ejection fraction decreased (Investigations) | 1 | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Bronchitis (Infections and infestations) | 3 | 1 | 1
Pyrexia (General disorders) | 1 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT04884191/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT04884191/SAP_001.pdf